CLINICAL TRIAL: NCT04558320
Title: COVID-19 and Lactating Mothers
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); New York University (Other)
Responsible Party: Principal Investigator, Kirsi Jarvinen-Seppo, Associate Professor, University of Rochester
Other Study IDs: STUDY00004889; 3U01AI131344-04S1 (NIH)
Record Dates: First submitted 2020-09-19; First posted 2020-09-22 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine if there may be COVID-19 virus in various samples collected from mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

* Currently lactating mother:

  * English-speaking
  * greater than or equal to 18 years of age
  * Assigned female at birth (AFAB)
  * Having a positive COVID-19 test within 14 days
* Child:

  * Infants younger than or equal to 6 months of age, exclusively or partially human milk fed, sourced from mother. Infants who are fed both directly at the breast and exclusively fed mother's milk via bottle will be included

Exclusion Criteria:

* Non-English speaking

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will include 50 adult lactating parents with COVID-19, and their infants (total sample size = 100). Participants can be residing anywhere in the continental United States.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
mean change in SARS-Cov-2 viral load in breast milk | baseline, days 3, 10, 19, 28 and 90
  RNA will be extracted from all sample types and SARS-CoV-2 primers used to amplify any present viral RNA using real-time qPCR. Repeated measures analysis will be used to compare the changes in sample viral load over time between women with mild to severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided